CLINICAL TRIAL: NCT01340092
Title: Use of a Family Navigator in Families With Children Newly Diagnosed With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Marilyn Augustyn, BMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 29964; HRSA R40MC19928-01-00 (Other Grant/Funding Number: HRSA)
Record Dates: First submitted 2011-04-20; First posted 2011-04-22 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Autistic Disorder
Keywords: Family Navigator; Autistic Disorder; Early Intervention; Developmental Disabilities; Child Development Disorders
MeSH Terms: conditions — Autistic Disorder; Developmental Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Navigator (Active Comparator): Family navigation
  Interventions: Other: Family Navigator
- Standard Care (No Intervention): standard care

INTERVENTIONS:
Other: Family Navigator — Families in the intervention group will receive approximately six sessions with a Family Navigator. The Family Navigator will:
  1. Help family identify key issues they need to address to get their child autism-specific services
  2. Help family address barriers to obtaining these services and strategize approaches to overcome them.
  Arms: Family Navigator

SUMMARY:
The purpose of this study is to see whether or not Family Navigators, who 1 ) help families after their child is diagnosed with autism and help them get autism specific services for their child 2) help families identify barriers to obtaining these services and 3) help families problem solve to overcome these barrier, are helpful to parents of a child newly diagnosed with an Autism Spectrum Disorder.

ELIGIBILITY:
Inclusion Criteria:

* Child with a new confirmed diagnosis of Autism Spectrum Disorder
* Child is under 8 years of age
* Parent is the mother, father and/or legal guardian of the child and identifies themselves as the primary caregiver
* Primary caregiver speaks English, Spanish, Haitian Creole, Somali, Vietnamese, Portuguese or Chinese

Exclusion Criteria:

* Parent or legal guardian has psychosis
* Parent or legal guardian endorses suicidal ideation
* Parent or legal guardian actively using illicit drugs
* Parent or legal guardian expected to leave area within 6 months

Ages: 15 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Actual)
Dates: Start 2011-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Hours of Services | 6 months after enrollment
  Mean number of autism-specific service hours received per week
Receipt of adequate services | 6 months after enrollment
  As defined by 25 hours/week
Time to Receipt of Services | 6 months after enrollment
  Difference between the date of the IEP/IFPS and date the child first received services

SECONDARY OUTCOMES:
Family Psychological Functioning | 6 months after enrollment
  * Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR).
  * Parenting Stress - Short Form (PSI)
  * Perceived Stress Scale- Self-Report (PSS)
  * Medical Outcomes Study Social Support (MOS-SS)
Family Psychological Functioning | Baseline
  * Quick Inventory of Depressive Symptomatology-Self Rated (QIDS-SR).
  * Parenting Stress - Short Form (PSI)
  * Perceived Stress Scale- Self-Report (PSS)
  * Medical Outcomes Study Social Support (MOS-SS)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Augustyn, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No